CLINICAL TRIAL: NCT01606631
Title: Evaluation of the Protective Role of Beta-blockers Prescribed in a Chronic Way on the Arisen of a Severe Septic Syndrome or a Toxic Shock at Patients Having a Community Infection
Brief Title: Role of Beta-blockers in the Prevention on the Arisen of a Severe Sepsis (TESS)
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CNIL AR091723
Record Dates: First submitted 2012-02-24; First posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-04

CONDITIONS: Community-Acquired Infections
Keywords: severe sepsis; toxic shock
MeSH Terms: conditions — Community-Acquired Infections; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Non applicable.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1 : experimental (case): Patients included in the study and admitted to the ICU either directly from UAA or after a hospitalization in a specialty, for a severe sepsis or septic shock on their infectious disease community.
- Arm 2 : control: Patients included in the study with an infectious disease community, admitted to a specialty, and have not progressed to severe sepsis or septic shock before hospital discharge.

SUMMARY:
The severe sepsis (SS) and toxic shock (TS) are both frequent and severe complications of infectious diseases. They are one of the top ten causes of death in industrialized countries. But an eventual protective role of beta-blockers (anti-hypertensive drug) in their occurrence on a community infection has never been studied. The objective of this study is to evaluate this role.

DETAILED DESCRIPTION:
The severe sepsis (SS) and toxic shock (TS) are both frequent and severe complications of infectious diseases. They are one of the top ten causes of death in industrialized countries. The adrenergic system is heavily involved in this pathological/physiological context. If the effect of various therapeutic strategies allowing the care of the SS/TS was widely estimated, the impact, positive or negative, therapeutic prescribed in the long term or more punctually - but be that as it may before the arisen of the sepsis - on the evolution of a community acute infectious pathology towards the SS/TS, had only little studied.

The main objective of this study is to estimate the possible protective role of a long-term prescription of a beta-blocker on the arisen of the SS/TS in patients having an acute infectious pathology of community origin.

The secondary objective will be to estimate, at the patients having developed a SS/TS, the impact of this long-term prescription of beta-blockers on the mortality in intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Common characteristics of cases and controls:
* Patients aged of more than 18 years old
* Hospitalized patients, during the period of study, via the ICU of the participating hospital center, for a community infectious pathology:

  * lower respiratory infections (pneumonia)
  * intra-abdominal infections (cholangitis, diverticulitis, peritonitis)
  * urinary parenchymal infection (pyelonephritis complicated or without abscess, prostatitis, orchitis, epididymitis)
  * infections of skin and soft tissue infections (cellulitis, fasciitis)
  * meningitis, endocarditis, osteo-articular infections, salpingitis

Definition of cases:

* Patient included in the study and admitted to the emergency service either directly from ICU or after a hospitalization in a specialty for severe sepsis or septic shock on their infectious disease community.

Definition of controls:

* Patient included in the study with an infectious disease community, admitted to a specialty, and have not progressed to severe sepsis or septic shock before being released from the hospital.

Non inclusion Criteria:

* Opposition of the patient to the IT processing of its data within the framework of this observational study.
* Exclusion criteria: Occurrence, during hospitalization, a severe sepsis or septic shock associated with a nosocomial superinfection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case : patients included in the study and admitted to the ICU either directly from UAA or after a hospitalization in a specialty, for a severe sepsis or septic shock on their infectious disease community.
  Control : patients included in the study with an infectious disease community, admitted to a specialty, and have not progressed to severe sepsis or septic shock before hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 2444 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the occurrence of severe sepsis, moving toward or away from septic shock. | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  From the date of randomization until the date of first documented assessed severe sepsis (moving toward or away from septic shock) up to the end of hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: Bellissant Eric, MD, PhD, Study Director — Rennes University Hospital - CIC
Locations (9):
- France (9):
  - Rennes University Hospital (Pontchaillou), Rennes, Ille-et-Vilaine
  - Brest University Hospital, Brest
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Groupe hospitalier Raymond Poincaré, AP-HP, Garches
  - Grenoble University Hospital (A. Michallon), Grenoble
  - Limoges University Hospital (Hospital Dupuytren), Limoges
  - Nancy University Hospital (Jeanne d'Arc), Nancy
  - Saint Etienne University Hospital (Bellevue), Saint-Etienne
  - Tours University Hospital (Bretonneau), Tours